CLINICAL TRIAL: NCT06470841
Title: CHG Regimen Combined With Venetoclax and Azacytidine in Newly Diagnosed Acute Myeloid Leukemia
Brief Title: CHG Combined With Venetoclax and Azacytidine in Newly Diagnosed AML
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liren Qian, Vice Director, Navy General Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WATCH2023
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHG Combined With Venetoclax and Azacytidine (Experimental): Patients were treated by CHG Combined With Venetoclax and Azacytidine
  Interventions: Drug: CHG Combined With Venetoclax and Azacytidine

INTERVENTIONS:
Drug: CHG Combined With Venetoclax and Azacytidine — Patients were treated by CHG Combined With Venetoclax and Azacytidine:
  Venetoclax 100mg po qd d1, 200mg po qd d2, 400mg po qd d3-14; Azacytidine 75 mg/m2 subcutaneous injection qd d1-7; Homoharringtonine 1mg/m2 iv qd d1-14; Cytarabine 10mg/m2 subcutaneous injection q12h d1-14; G 250ug/m2 subcutaneous injection qd d0-14.
  Other Names: VACHG

SUMMARY:
The goal of this phase 2 trial is to test the safety and efficacy of CHG Combined With Venetoclax in treating patients with newly diagnosed AML.

DETAILED DESCRIPTION:
The investigators will evaluate response rate of CHG regimen Combined With Venetoclax in newly diagnosed acute myeloid leukemia. After induction therapy, patients will be given standardized treatment according to risk stratification according to NCCN guidelines. Progression free survival (PFS), Overall survival (OS), and Toxicity will be counted.

ELIGIBILITY:
Inclusion Criteria:

* The patient should, in the investigator's opinion, be able to meet all clinical trial requirements.
* The patient is willing and able to adhere to the study visit schedule and other protocol requirements.
* The patient should be diagnosed with AML according to the standard criteria of the World Health Organisation (WHO).
* The patient should not have received any prior treatment for AML.

Exclusion Criteria:

* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment.
* Any instability of systemic disease, including but not limited to severe cardiac, liver, kidney, or metabolic disease need therapy.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  ORR was defined as the proportion of patients who achieved CR or PR as their best response

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 3 years
  OS was defined as time from diagnosis to death from any cause or the last follow-up
Progression Free Survival (PFS) | 2 years
  For patients in morphologic remission, documented relapse was considered progression. Relapse following complete remission(CR) is defined as reappearance of leukemic blasts in the peripheral blood or the finding of more than 5% blasts in the BM, not attributable to another cause (eg, BM regeneration after consolidation therapy) or extramedullary relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Liren Qian, PhD, Principal Investigator — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China